CLINICAL TRIAL: NCT00581737
Title: Cognitive Functioning and Quality of Life in CNS Lymphoma
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00-083
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma; Central Nervous System Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

SUMMARY:
The purpose of this study is to evaluate several aspects of thinking abilities including attention and memory, and quality of life in patients who were diagnosed with and treated for Primary CNS Lymphoma (PCNSL), and are in remission of their disease. The findings of this study may help us understand whether this disease and its treatment may have affected some patients' thinking skills, and may provide important information that can be used to develop programs to improve the quality of life of patients with PCNSL.

This research will also study whether persons having particular types of genes involved in the metabolism of methionine (5-methyltetrahydrofolate-homocysteine S-methyltransferase-MTR, MTFH reductase-MTFHR, transcobalamin 2-Tc2), and apolipoprotein E (APOE) are more likely to have delayed adverse effects after treatment for their tumors. The findings of this study may help us understand whether this disease and its treatment may have affected some patients' thinking skills, and whether this may be related to having certain genes.

DETAILED DESCRIPTION:
The incidence of primary central nervous system lymphoma (PCNSL) has increased threefold in immunocompetent populations in recent years. Improvements in treatment, particularly involving combined modality therapy with chemotherapy and radiotherapy have been shown to augment patient survival with a median disease-free period of about 40 months. However, the combination of these two modalities often increases the risk for delayed neurotoxicity. There is a paucity of studies that have assessed neuropsychological functioning and quality of life in patients with PCNSL. The majority of studies reported performance status and survival rates, but systematic cognitive evaluations were only seldom included. Unfortunately, relying only on these variables does not adequately assess the more subtle cognitive impairments that most patients with brain tumors experience. Neuropsychological difficulties often interfere with disease free patients' ability to function at premorbid levels at work and at home. A study including neuropsychological evaluations of a relatively large group of patients with PCNSL who received combined modality treatments, and are in remission from their disease is planned. A follow-up assessment also will be performed in order to monitor performance over a specified period of time. The proposed study will also test the hypotheses that: (1) the presence of polymorphisms that influence methionine metabolism places PCNSL patients treated with chemotherapy alone or in combination with radiotherapy at risk for developing treatment-induced white matter disease and cognitive dysfunction; (2) the possession of the apolipoprotein E (APOE) є-4 allele is associated with the development of cognitive difficulties following treatment for PCNSL. Research in order to better understand the incidence, extent, and severity of treatment-induced neuropsychological impairments in patients with PCNSL is of utmost importance, given the recent increase in both the number of cases diagnosed and longterm survival. It is likely to provide valuable information regarding specific cognitive domains that should be addressed in the development of strategies for cognitive rehabilitation or other interventions that may be appropriate. The findings of this study will also be relevant for comparison with ongoing and future research investigating the potential neurocognitive sequelae of alternative treatment modalities for PCNSL (e.g., high-dose chemotherapy followed by peripheral blood progenitor cell (PBPC) transplant).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of and treatment for PCNSL
* Disease in remission at the time of testing, as defined by negative MRI and/or CSF cytology, and ocular exam if initially positive
* English speaking

Exclusion Criteria:

* patients who are medically unstable
* patients with severe, decompensated psychiatric disorders
* patients with a pre-existing neurological condition other than the designated illness (e. g., head trauma)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2000-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The goal of this study is to examine the neurobehavioral functioning of PCNSL survivors who received radiation and chemotherapy treatments, and are in remission from their disease. | 2 years

SECONDARY OUTCOMES:
Examine the delayed effects of whole-brain radiation and chemotherapy on several aspects of cognitive functioning, and quality of life. Also, perform a follow-up evaluation in order to monitor neurocognitive functioning over a specified period of time. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Denise Correa, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org